CLINICAL TRIAL: NCT02688842
Title: The Safety and Effectiveness Evaluation of New Specifications (38mm) of FirehawkTM Sirolimus Target-eluting Coronary Stent System in the Treatment of Coronary Heart Disease: a Prospective, Multicenter, Single-group Study.
Brief Title: Evaluation of New Specifications (38mm) of FirehawkTM in the Treatment of Coronary Heart Disease
Acronym: Firehawk_38
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai MicroPort Medical (Group) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Firehawk_LS
Record Dates: First submitted 2016-02-18; First posted 2016-02-23 (Estimated); Results first posted 2020-02-20 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2021-05

CONDITIONS: Coronary Heart Disease
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Intervention Model Description: all patients implanted Firehawk stent of new specification (38mm long)
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- treatment group (Experimental): Implantation of the released specification (38mm) of FirehawkTM rapamycin target-eluting coronary stent systems
  Interventions: Device: Rapamycin target-eluting coronary stent systems (38mm)

INTERVENTIONS:
Device: Rapamycin target-eluting coronary stent systems (38mm)
  Other Names: Firehawk-38

SUMMARY:
The purpose of this study is to evalute the clinical safety and effectiveness of released specification (38mm) of FirehawkTM Sirolimus target-eluting coronary stent system.

ELIGIBILITY:
Inclusion Criteria:

1. 18-80 years of age, males or non-pregnant women;
2. Evidence of silent ischemia, stability or in patients with old myocardial infarction or unstable angina;
3. Primary target lesion, in situ coronary artery disease;
4. Target lesion length ≤ 60mm, target lesion diameter 2.75mm or 4.0mm (Visual method);
5. The target lesion diameter stenosis ≥ 70% (Visual method);
6. Each target lesion implantation the same stent (Firehawk stand);
7. With indications for coronary artery bypass surgery;
8. To understand the purpose of testing, voluntary and informed consent, patients undergoing invasive imaging follow-up.

Exclusion Criteria:

1. Within 72h of any acute myocardial infarction;
2. Unprotected left main coronary artery disease, triple vessel lesions which need treated all;
3. Severe calcified lesions that cannot be successfully expanded and distorting lesions not suitable for stent delivery;
4. Artery and/or vein bypass graft lesions;
5. Intracoronary implantation of any branding stents within 1 year;
6. Severe congestive heart failure (NYHA class III and above), or left ventricular ejection fraction <35% (ultrasound or left ventricular angiography);
7. Preoperative renal function serum creatinine >2.0mg/DL;
8. Bleeding, active gastrointestinal ulcers, brain hemorrhage or subarachnoid hemorrhage and half year history of ischemic stroke, antiplatelet agents and would not allow an anticoagulant therapy contraindications patients undergoing antithrombotic therapy;
9. Aspirin, clopidogrel, heparin, contrast agent, poly lactic acid polymer and rapamycin allergies;
10. The patient's life expectancy is less than 12 months;
11. Top participated in other drug or medical device and does not meet the primary study endpoint in clinical trials time frame;
12. Researchers determine patient compliance is poor, unable to complete the study in accordance with the requirements;
13. Heart transplantation patients.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2021-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Runlin Gao, MD, Principal Investigator — Fu Wai Hospital & National Center for Cardiovascular Diseases in China
Locations (1):
- Fu Wai Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Group: Implantation of the released specification (38mm) of FirehawkTM rapamycin target-eluting coronary stent systems
  Rapamycin target-eluting coronary stent systems (38mm)
Period: Overall Study
Arm/Group | Treatment Group
Started | 38
Completed | 38
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment Group
Number analyzed (Participants) | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (9.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 30
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  China | 38
Diabetes Mellitus (DM) history [Count of Participants; unit: Participants]
  With DM | 13
  Without DM | 25
Coronary Artery Disease (CAD) history [Count of Participants; unit: Participants]
  With CAD | 7
  Without CAD | 31
hypertension (HTN) history [Count of Participants; unit: Participants]
  With HTN | 27
  Without HTN | 11
Cigarette usage [Count of Participants; unit: Participants]
  Never | 17
  Smoker | 15
  Quit smoking | 1
  Relapse | 5
Myocardial Infarction (MI) history [Count of Participants; unit: Participants]
  With MI | 13
  Without MI | 25

OUTCOME MEASURES:

1. Primary Outcome: In-stent Late Lumen Loss
Time Frame: 9 month after stent implantation
Population: A sum of 31 patients with 33 target lesions were analyzed by Quantitative Coronary Angiography (QCA). 7 participants did not participate in 9 month angiographic follow up.
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: target stent
Arm/Group | Treatment Group
Number analyzed (Participants) | 31
Number analyzed (target stent) | 33
mm | 0.19 (0.43)

2. Secondary Outcome: Participants With Target Lesion Failure
Description: a composite endpoint of cardiac death, myocardial infarction related to target vessel (TVMI) and clinically-indicated revascularization related to target lesion (CI-TLR)
Time Frame: 30 days after stent implantation
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group
Number analyzed (Participants) | 38
Participants | 1

3. Secondary Outcome: Participants With Target Lesion Failure
Description: as for outcome 2
Time Frame: 6months after stent implantation
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group
Number analyzed (Participants) | 38
Participants | 1

4. Secondary Outcome: Participants With Target Lesion Failure
Description: as for outcome 2
Time Frame: 12 months after stent implantation
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group
Number analyzed (Participants) | 38
Participants | 2

5. Secondary Outcome: Participants With Target Lesion Failure
Description: as for outcome 2
Time Frame: 2 years after stent implantation
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group
Number analyzed (Participants) | 38
Participants | 2

6. Secondary Outcome: Participants With Target Lesion Failure
Description: as for outcome 2
Time Frame: 3 years after stent implantation
Population: One participant was lost during 3 years follow up.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group
Number analyzed (Participants) | 37
Participants | 2

7. Secondary Outcome: Participants With Target Lesion Failure
Description: as for outcome 2
Time Frame: 4 years after stent implantation
Population: One participant was lost during 4 years follow up.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group
Number analyzed (Participants) | 37
Participants | 2

8. Secondary Outcome: Major Adverse Cardiac Events
Description: composite endpoint of all cause death, any myocardial infarction and any revascularization
Time Frame: 30 days after stent implantation
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group
Number analyzed (Participants) | 38
Participants | 1

9. Secondary Outcome: Major Adverse Cardiac Events
Description: composite endpoint of all cause death, any myocardial infarction and any revascularization
Time Frame: 6 months after stent implantation
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group
Number analyzed (Participants) | 38
Participants | 1

10. Secondary Outcome: Major Adverse Cardiac Events
Description: composite endpoint of all cause death, any myocardial infarction and any revascularization
Time Frame: 12 months after stent implantation
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group
Number analyzed (Participants) | 38
Participants | 4

11. Secondary Outcome: Major Adverse Cardiac Events
Description: composite endpoint of all cause death, any myocardial infarction and any revascularization
Time Frame: 2 years after stent implantation
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group
Number analyzed (Participants) | 38
Participants | 5

12. Secondary Outcome: Major Adverse Cardiac Events
Description: composite endpoint of all cause death, any myocardial infarction and any revascularization
Time Frame: 3 years after stent implantation
Population: One participant was lost during 3 years follow up.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group
Number analyzed (Participants) | 37
Participants | 6

13. Secondary Outcome: Major Adverse Cardiac Events
Description: composite endpoint of all cause death, any myocardial infarction and any revascularization
Time Frame: 4 years after stent implantation
Population: One participant was lost during 4 years follow up.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group
Number analyzed (Participants) | 37
Participants | 7

ADVERSE EVENTS:
Time Frame: 4 year follow up
Arm/Group | Treatment Group
All-Cause Mortality (participants affected / at risk) | 0/38
Serious Adverse Events (participants affected / at risk) | 15/38
Other Adverse Events (participants affected / at risk) | 25/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group (N=38)
Target Lesion Revascularization (Cardiac disorders) | 1 (1)
Angina (Cardiac disorders) | 5 (5)
Rehospitalization (General disorders) | 8 (8)
lymphoma (Blood and lymphatic system disorders) | 1 (1)
myocardial infarction (Cardiac disorders) | 2 (2)
non-Target Vessel Revascularization (Cardiac disorders) | 4 (4)
acute cerebral infarction (Nervous system disorders) | 1 (1)
Diastolic dysfunction (Cardiac disorders) | 1 (1)
gastric antrum erosion (Gastrointestinal disorders) | 1 (1)
senile cataract (Eye disorders) | 2 (2)
coronary artery disease (Cardiac disorders) | 1 (1)
Diabetes Mellitus (Metabolism and nutrition disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group (N=38)
elevated myocardial enzyme (Cardiac disorders) | 2 (2)
corneal ulcer (Eye disorders) | 1 (1)
hypokalemia (General disorders) | 1 (1)
aneurysm (Vascular disorders) | 1 (1)
atrial fibrillation (Cardiac disorders) | 1 (1)
Infection (Infections and infestations) | 5 (5)
heart discomfort after movation (Cardiac disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chronic gastroenteritis (Gastrointestinal disorders) | 1 (1)
Short breath (Respiratory, thoracic and mediastinal disorders) | 1 (1)
renal cyst (Renal and urinary disorders) | 1 (1)
premature ventricular contraction (Cardiac disorders) | 1 (1)
myocardial injury (Cardiac disorders) | 13 (13)
Pain (General disorders) | 1 (1)
vertigo (Nervous system disorders) | 1 (1)
palpitation (Cardiac disorders) | 1 (1)
angina (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No